CLINICAL TRIAL: NCT01574209
Title: Gut Peptides and Intestinal Permeability in Celiac Patients, Healthy Subjects and IBS Patients: a Comparative Study
Brief Title: Gut Peptides and Intestinal Permeability in Celiac Disease and Irritable Bowel Syndrome
Acronym: PPCD
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Giuseppe Riezzo, Director of Experimental Pathophysiology Laboratory, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Other Study IDs: CD5X1000
Record Dates: First submitted 2012-03-28; First posted 2012-04-10 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Celiac Disease; Irritable Bowel Syndrome
Keywords: Celiac disease; IBS; Intestinal barrier; Intestinal permeability; GI peptides
MeSH Terms: conditions — Celiac Disease; Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Celiac Disease: Patients suffering from coeliac diseases confirmed by small intestinal biopsy
- IBS patients: Patients suffering from irritable bowel syndrome (IBS) according to Rome III criteria
- Healthy subjects: Healthy subjects as control group

SUMMARY:
It is well known that the intestinal barrier is altered in celiac disease (CD), an autoimmune disease that develops in genetically predisposed subjects exposed to ingestion of wheat gliadin and of related prolamines of barley and rye. More recently, defective epithelial barrier has been implicated in the pathogenesis of other conditions such as irritable bowel syndrome (IBS). At present IBS is still considered a functional condition although low-grade inflammation has been associated with its manifestation, particularly that following infection. Different substances have been implicated in the (dis)regulation of intestinal barrier, among them zonulin seems to play a key role. Other gastrointestinal peptides are GPL-2, Ghrelin, and Epidermal growth factor (EGF). In order to shed light on the hormonal regulation of intestinal barrier function in celiac patients before undergoing a gluten free diet and possible differences with those of IBS patients, in the present study the investigators will apply the non-invasive lactulose/mannitol permeability test toward the evaluation of intestinal damage. The pattern of intestinal permeability and the GI peptides concentration will be compared in celiac patients, IBS patients and healthy controls.

ELIGIBILITY:
Inclusion criteria of celiac disease patients:

* Diagnosis of CD was based on the detection of IgA antiendomysial and IgA antitissue transglutaminase antibodies in serum
* Diagnosis must be confirmed by a small intestinal biopsy obtained at the time of gastrointestinal endoscopy.
* All patients must show Marsh 3 grade villous atrophy at the time of the diagnosis.

Inclusion criteria of IBS patients.

* Subjects suffering from irritable bowel syndrome according to the Rome III criteria.
* Availability of at least one GI imaging study during the last five years (colonoscopy, sigmoidoscopy, abdominal ultrasound, barium enema)

Exclusion criteria for both the above groups:

* None were taking anti-inflammatory drugs (including mast cell stabilisers, histamine antagonists, anticholinergics, anti-diarrhoea medication, probiotics, immunosuppressants and steroids)
* Presence of organic syndrome, including food allergy, atopy and severe clinical depression or anxiety.
* Abnormal laboratory data or thyroid function
* Major abdominal surgery Healthy subjects will be recruited in the administrative staff of the Institute after thorough exclusion of GI symptoms.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatients recruited in IRCCS "S. de Bellis"
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2012-04; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of GI peptides (Zonulin, GLP-2, Ghrelin and EGF) | within one month after the enrollment

SECONDARY OUTCOMES:
Intestinal permeability | within one month after the enrollment
  The detection and measurement of two sugar probes, lactulose (La) and mannitol (Ma), in the urine will be performed by chromatographic analysis. For each sample the percentage of ingested La and Ma in urine will be evaluated and their ratio (La-Ma) will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Riezzo, MD, Principal Investigator — National Institute of Digestive Diseases IRCCS "S. de Bellis"
Locations (1):
- National Institute of Digestive Diseases IRCCS "S. de Bellis", Castellana Grotte, Bari, Italy

REFERENCES:
- [Background] Fasano A. Zonulin and its regulation of intestinal barrier function: the biological door to inflammation, autoimmunity, and cancer. Physiol Rev. 2011 Jan;91(1):151-75. doi: 10.1152/physrev.00003.2008. PMID 21248165
- [Background] Cani PD, Possemiers S, Van de Wiele T, Guiot Y, Everard A, Rottier O, Geurts L, Naslain D, Neyrinck A, Lambert DM, Muccioli GG, Delzenne NM. Changes in gut microbiota control inflammation in obese mice through a mechanism involving GLP-2-driven improvement of gut permeability. Gut. 2009 Aug;58(8):1091-103. doi: 10.1136/gut.2008.165886. Epub 2009 Feb 24. PMID 19240062
- [Background] Gecse K, Roka R, Sera T, Rosztoczy A, Annahazi A, Izbeki F, Nagy F, Molnar T, Szepes Z, Pavics L, Bueno L, Wittmann T. Leaky gut in patients with diarrhea-predominant irritable bowel syndrome and inactive ulcerative colitis. Digestion. 2012;85(1):40-6. doi: 10.1159/000333083. Epub 2011 Dec 14. PMID 22179430
- [Background] Menard S, Lebreton C, Schumann M, Matysiak-Budnik T, Dugave C, Bouhnik Y, Malamut G, Cellier C, Allez M, Crenn P, Schulzke JD, Cerf-Bensussan N, Heyman M. Paracellular versus transcellular intestinal permeability to gliadin peptides in active celiac disease. Am J Pathol. 2012 Feb;180(2):608-15. doi: 10.1016/j.ajpath.2011.10.019. Epub 2011 Nov 24. PMID 22119716
- [Background] Malandrino N, Capristo E, Farnetti S, Leggio L, Abenavoli L, Addolorato G, Gasbarrini G. Metabolic and nutritional features in adult celiac patients. Dig Dis. 2008;26(2):128-33. doi: 10.1159/000116770. Epub 2008 Apr 21. PMID 18431062
- [Derived] Linsalata M, Riezzo G, D'Attoma B, Clemente C, Orlando A, Russo F. Noninvasive biomarkers of gut barrier function identify two subtypes of patients suffering from diarrhoea predominant-IBS: a case-control study. BMC Gastroenterol. 2018 Nov 6;18(1):167. doi: 10.1186/s12876-018-0888-6. PMID 30400824
- [Derived] Russo F, Chimienti G, Clemente C, D'Attoma B, Linsalata M, Orlando A, De Carne M, Cariola F, Semeraro FP, Pepe G, Riezzo G. Adipokine profile in celiac patients: differences in comparison with patients suffering from diarrhea-predominant IBS and healthy subjects. Scand J Gastroenterol. 2013 Dec;48(12):1377-85. doi: 10.3109/00365521.2013.845907. Epub 2013 Oct 28. PMID 24164320